CLINICAL TRIAL: NCT04199468
Title: An Electrophysiological Examination of CB1 and NMDA Receptors in Humans
Brief Title: THC and Ketamine Effects in Humans: Relation to Neural Oscillations and Psychosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Rajiv Radhakrishnan, MD, Assistant Professor, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2000025927; 000 (Other: CTGTY)
Record Dates: First submitted 2019-10-21; First posted 2019-12-16 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Cannabis; Ketamine
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Active Delta-9-THC and Placebo Ketamine (Experimental): Active IV Delta-9-THC and Placebo Ketamine
  Interventions: Drug: Active Delta-9-THC; Drug: Placebo Ketamine
- Active Delta-9-THC and Active Ketamine (Experimental): Active IV Delta-9-THC and Active Ketamine
  Interventions: Drug: Active Delta-9-THC; Drug: Active Ketamine
- Placebo Delta-9-THC and Placebo Ketamine (Experimental): IV Placebo Delta-9-THC and Placebo Ketamine
  Interventions: Drug: Placebo Delta-9-THC; Drug: Placebo Ketamine
- Placebo Delta-9-THC and Active Ketamine (Experimental): IV Placebo Delta-9-THC and Active Ketamine
  Interventions: Drug: Placebo Delta-9-THC; Drug: Active Ketamine

INTERVENTIONS:
Drug: Active Delta-9-THC — Active Delta-9-THC (0.015 mg/kg) given intravenously (IV)
  Arms: Active Delta-9-THC and Active Ketamine; Active Delta-9-THC and Placebo Ketamine
Drug: Placebo Delta-9-THC — A placebo dose given intravenously (IV)
  Arms: Placebo Delta-9-THC and Active Ketamine; Placebo Delta-9-THC and Placebo Ketamine
Drug: Active Ketamine — Active Ketamine (0.2 mg/kg) given intravenously (IV)
  Arms: Active Delta-9-THC and Active Ketamine; Placebo Delta-9-THC and Active Ketamine
Drug: Placebo Ketamine — A placebo dose given intravenously (IV)
  Arms: Active Delta-9-THC and Placebo Ketamine; Placebo Delta-9-THC and Placebo Ketamine

SUMMARY:
The aim of the research protocol is to evaluate cannabinoid-glutamate interactions in humans. As part of this aim the investigators will assess the safety and tolerability of the combination of NMDA antagonist, ketamine, and the cannabinoid, delta-9-tetrahydrocannabinol (THC), in healthy adult subjects, and characterize the interactive effects of ketamine and THC on various electrophysiological (EEG), cognitive, and behavioral outcomes.

DETAILED DESCRIPTION:
The investigators will examine the contributions of the cannabinoid receptor (CB1R) and N-methyl D-aspartate receptor (NMDAR) systems to psychosis in healthy humans beings using THC and ketamine respectively (both alone and in combination). Healthy subjects (n=21) will receive THC (active or placebo) followed by ketamine (active or placebo) in a double blind, randomized, crossover (2x2) design. Psychotomimetic effects will be assessed before and at various time points after the drug infusions. EEG indices of information processing, specifically neural oscillations, will be assessed during peak drug effects.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to approximately 45 years old
2. Good physical and mental health as determined by history, the Structured Clinical Interview for DSM-5 TR (SCID-NP) and collateral information, physical and laboratory examinations, ECG and vital signs.
3. Weight of 100 kg (220.46 lbs.) or less (inclusive).

Exclusion Criteria:

1. Unstable serious medical conditions. At the discretion of the investigator, subjects with unstable medical conditions that may necessitate changes in medical treatment and hence influence study outcomes will be excluded.
2. Uncontrolled hypertension, long QT syndrome, and seriously abnormal EKG results. EKG abnormalities will be reviewed by the PI and eligibility decisions will be made at the discretion of the PI.
3. A hearing deficit in greater than one band in an ear detected using a Welch-Allyn audioscope (500, 1000, 2000 and 4000 Hz threshold will be evaluated)
4. Positive pregnancy test

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
EEG Measures 1 | 0-60 minutes after the onset of drug infusion
  The primary EEG outcome 1 will be EEG event related potential voltage amplitude (microvolts).
EEG Measures 2 | 0-60 minutes after the onset of drug infusion
  The primary EEG outcome 2 will be EEG event related potential latency (milliseconds).
EEG Measures 3 | 0-60 minutes after the onset of drug infusion
  The primary EEG outcome 3 will be spectral power (microvolts squared).
EEG Measures 4 | 0-60 minutes after the onset of drug infusion
  The primary EEG outcome 4 will be Intertrial Coherence (phase locking factor).
EEG Measures 5 | 0-60 minutes after the onset of drug infusion
  The primary EEG outcome 5 will be neural noise (Lempel Ziv Complexity).
Neurochemical Measures: THC levels | -30, +25, +60, +120 minutes after start of drug infusion (0)
  THC blood levels (ng/mL) will be assayed to determine the relationships between blood levels and EEG measures (outcomes 1-5) and behavioral measures (outcomes 10-12). Blood sampled at 4 time-points will be centrifuged and the resultant plasma will be aliquoted into appropriate vials and stored at -80 degrees C until the time of the assay.
Neurochemical Measures: THC-COOH levels | -30, +25, +60, +120 minutes after start of drug infusion (0)
  THC-COOH blood levels (ng/mL) will be assayed to determine the relationships between blood levels and EEG measures (outcomes 1-5) and behavioral measures (outcomes 10-12). Blood sampled at 4 time-points will be centrifuged and the resultant plasma will be aliquoted into appropriate vials and stored at -80 degrees C until the time of the assay.
Neurochemical Measures: ketamine/norketamine levels | -30, +25, +60, +120 minutes after start of drug infusion (0)
  Ketamine/norketamine blood levels (ng/mL) will be assayed to determine the relationships between blood levels and EEG measures (outcomes 1-5) and behavioral measures (outcomes 10-12). Blood sampled at 4 time-points will be centrifuged and the resultant plasma will be aliquoted into appropriate vials and stored at -80 degrees C until the time of the assay.
Genetics | Collected at the screening visit.
  Blood samples for DNA extraction will be collected to examine whether any of the genes e.g., calcyon, BDNF, neuregulin-1, dysbindin, NOTCH4, COMT and the 22q11 PRODH2/DGCR6 locus that have been associated with schizophrenia, modify the effects of delta-9-THC, ketamine or the combination.

SECONDARY OUTCOMES:
Positive and Negative Symptoms Scale (PANSS) | -60, +70, +120, +240 from baseline (0) (units in minutes).
  Positive, negative, and general psychosis symptoms will be assessed using the Positive and Negative Syndrome Scale (PANSS). The PANSS is divided into three sub-scales: Positive Scale (7 items), Negative Scale (7 items), and General Psychopathology Scale (16 items). Each item is scored from 1 to 7 (1=absent, 2=minimum, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme). Scores range from 30 to 210, where higher scores indicate greater symptom severity.
Perceptual Alterations | -60, +70, +120, +240 from baseline (0) (units in minutes).
  Perceptual alterations will be measured using the Clinician Administered Dissociative Symptoms Scale (CADSS), a scale consisting of 19 self-report items and 8 clinician-rated items (0 = not at all, 4 = extremely) that we have shown to be sensitive to THC effects. The scale captures alterations in environmental/time/body perception, feelings of unreality, and memory impairment.
Cannabis Subjective Effects | -60, +70, +120, +240 from baseline (0) (units in minutes).
  Feeling states associated with cannabis intoxication will be measured using a self-reported visual analog scale of 3 feeling states ("high", "calm and relaxed", and "tired") associated with cannabis effects. Subjects will be asked to score the perceived intensity of these feeling states at that moment on a 100 mm line (0 = not at all, 100 = extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Radhakrishnan, M.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States